CLINICAL TRIAL: NCT00414934
Title: The Effectiveness of Whole-body 18F-NaF PET in Detecting Metastatic Bone Lesion for Patients With Cancer: A Comparison Study With 99mTc-MDP Bone Scintigraphy.
Brief Title: 18F-NaF PET in Detecting Metastatic Bone Lesion for Patients With Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Yen RF, National Taiwan University Hospital
Other Study IDs: 941220
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2009-08-17 (Estimated); Status verified 2009-08

CONDITIONS: Cancer
Keywords: cancer; bone scan; NaF bone PET
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- metastatic bone lesion for patients with cancer

SUMMARY:
18F ion is a positron emitting bone radiopharmaceuticals. The skeletal uptake of 18F relies on the exchange of hydroxyl ions in the hydroxyapatit crystal which is an indicator of bone metabolic activity (8). It has good soft tissue clearance and high affinity of to the bone matrix. It is able to perform a highly sensitive whole-body screening for bone metastases using a high resolution PET scanner. Therefore, we conduct a prospective study to evaluate the accuracy and clinical value of 18F PET in staging bone metastases by

1. Comparing the sensitivity of 18F-NaF PET with that of 99mTc-MDP scintigraphy;
2. Determining the clinical impact of PET results on subsequent patient management.

DETAILED DESCRIPTION:
Skeletal metastases are the most common cause of morbidity and mortality in patients with malignancy, especially in patients with breast cancer, lung cancer, prostate cancer and head & neck cancer. In patients with lung cancer, bone metastases are present in 20-30% of patient at initial diagnosis (1-2). Accuracy staging bone metastases can lead to modification of following treatment and evaluation of prognosis.

The planar whole-body 99mTc-methylene diphosphonate (MDP) radionuclide bone scintigraphy is the most widely used technique in detecting metastatic bone lesions at present. Abnormal tracer accumulation may occur at any skeletal site with an elevated rate of bone turnover. However, conventional planar bone scintigraphy was reported to be less sensitive than MRI in detecting spinal metastases (3-7).

18F ion is a positron emitting bone radiopharmaceuticals. The skeletal uptake of 18F relies on the exchange of hydroxyl ions in the hydroxyapatit crystal which is an indicator of bone metabolic activity (8). It has good soft tissue clearance and high affinity of to the bone matrix. It is able to perform a highly sensitive whole-body screening for bone metastases using a high resolution PET scanner.

To the best of our knowledge, there are only limited studies evaluating the clinical utilization of 18F-NaF PET for detection of bone metastases (10-12). Therefore, we would like to conduct a prospective study to evaluate the accuracy and clinical value of 18F PET in staging bone metastases by

1. Comparing the sensitivity of 18F-NaF PET with that of 99mTc-MDP scintigraphy;
2. Determining the clinical impact of PET results on subsequent patient management.

99mTc-MDP scintigraphy and 18F PET will be performed in 2 weeks for all patients. Interpretation of 99mTc-MDP scintigraphy and 18F PET will be performed following the criteria described by Crasnow et all (13). The accuracy of 99mTc-MDP scintigraphy and 18F PET detection of bone metastases for each patient will be determined by the histopathological results, MRI results, or other clinical evidences afterward.

ELIGIBILITY:
Inclusion Criteria:

* pathology proofed lung cancer and are referred to perform whole-body bone scintigraphies for staging metastatic bone diseases

Exclusion Criteria:

* patients whose age are below 18
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic bone lesion for patients with cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-10; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruoh-Fang Yen, M.D.,Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Tritz DB, Doll DC, Ringenberg QS, Anderson S, Madsen R, Perry MC, Yarbro JW. Bone marrow involvement in small cell lung cancer. Clinical significance and correlation with routine laboratory variables. Cancer. 1989 Feb 15;63(4):763-6. doi: 10.1002/1097-0142(19890215)63:43.0.co;2-f. PMID 2536586
- [Background] Bezwoda WR, Lewis D, Livini N. Bone marrow involvement in anaplastic small cell lung cancer. Diagnosis, hematologic features, and prognostic implications. Cancer. 1986 Oct 15;58(8):1762-5. doi: 10.1002/1097-0142(19861015)58:83.0.co;2-v. PMID 3019512
- [Background] Avrahami E, Tadmor R, Dally O, Hadar H. Early MR demonstration of spinal metastases in patients with normal radiographs and CT and radionuclide bone scans. J Comput Assist Tomogr. 1989 Jul-Aug;13(4):598-602. doi: 10.1097/00004728-198907000-00008. PMID 2745777
- [Background] Brown B, Laorr A, Greenspan A, Stadalnik R. Negative bone scintigraphy with diffuse osteoblastic breast carcinoma metastases. Clin Nucl Med. 1994 Mar;19(3):194-6. doi: 10.1097/00003072-199403000-00005. PMID 8033466
- [Background] Thrupkaew AK, Henkin RE, Quinn JL 3rd. False negative bone scans in disseminated metastatic disease. Radiology. 1974 Nov;113(2):383-6. doi: 10.1148/113.2.383. No abstract available. PMID 4419062
- [Background] Haubold-Reuter BG, Duewell S, Schilcher BR, Marincek B, von Schulthess GK. The value of bone scintigraphy, bone marrow scintigraphy and fast spin-echo magnetic resonance imaging in staging of patients with malignant solid tumours: a prospective study. Eur J Nucl Med. 1993 Nov;20(11):1063-9. doi: 10.1007/BF00173484. PMID 8287874
- [Background] Frank JA, Ling A, Patronas NJ, Carrasquillo JA, Horvath K, Hickey AM, Dwyer AJ. Detection of malignant bone tumors: MR imaging vs scintigraphy. AJR Am J Roentgenol. 1990 Nov;155(5):1043-8. doi: 10.2214/ajr.155.5.2120933.
- [Background] Hawkins RA, Choi Y, Huang SC, Hoh CK, Dahlbom M, Schiepers C, Satyamurthy N, Barrio JR, Phelps ME. Evaluation of the skeletal kinetics of fluorine-18-fluoride ion with PET. J Nucl Med. 1992 May;33(5):633-42. PMID 1569473
- [Background] Schirrmeister H, Guhlmann A, Kotzerke J, Santjohanser C, Kuhn T, Kreienberg R, Messer P, Nussle K, Elsner K, Glatting G, Trager H, Neumaier B, Diederichs C, Reske SN. Early detection and accurate description of extent of metastatic bone disease in breast cancer with fluoride ion and positron emission tomography. J Clin Oncol. 1999 Aug;17(8):2381-9. doi: 10.1200/JCO.1999.17.8.2381. PMID 10561300
- [Background] Schirrmeister H, Guhlmann A, Elsner K, Kotzerke J, Glatting G, Rentschler M, Neumaier B, Trager H, Nussle K, Reske SN. Sensitivity in detecting osseous lesions depends on anatomic localization: planar bone scintigraphy versus 18F PET. J Nucl Med. 1999 Oct;40(10):1623-9. PMID 10520701
- [Background] Schirrmeister H, Glatting G, Hetzel J, Nussle K, Arslandemir C, Buck AK, Dziuk K, Gabelmann A, Reske SN, Hetzel M. Prospective evaluation of the clinical value of planar bone scans, SPECT, and (18)F-labeled NaF PET in newly diagnosed lung cancer. J Nucl Med. 2001 Dec;42(12):1800-4. PMID 11752076
- [Background] Hetzel M, Arslandemir C, Konig HH, Buck AK, Nussle K, Glatting G, Gabelmann A, Hetzel J, Hombach V, Schirrmeister H. F-18 NaF PET for detection of bone metastases in lung cancer: accuracy, cost-effectiveness, and impact on patient management. J Bone Miner Res. 2003 Dec;18(12):2206-14. doi: 10.1359/jbmr.2003.18.12.2206. PMID 14672356
- [Background] Krasnow AZ, Hellman RS, Timins ME, Collier BD, Anderson T, Isitman AT. Diagnostic bone scanning in oncology. Semin Nucl Med. 1997 Apr;27(2):107-41. doi: 10.1016/s0001-2998(97)80043-8. PMID 9144855